CLINICAL TRIAL: NCT05772897
Title: Effects of Attachment-Focused Parenting Intervention on Postpartum Depression and Biological Markers of Stress in Mothers and Their Infants
Brief Title: Parenting Skills Group for Mothers With Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-2593
Record Dates: First submitted 2023-02-08; First posted 2023-03-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: All participants will ultimately receive the parenting group intervention. A waitlist control design will be implemented to compare outcomes between those not having received the intervention yet and those having completed it. Data collection will occur pre-intervention, immediately post-intervention, at 6 months post-intervention, at 12 months post-intervention, and at approximately 5 years post-intervention (when child is school-aged).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circle of Security Parenting (COSP) group (Experimental): This group of mothers will be assigned to begin the parenting skills intervention (COSP) group soon after enrollment, and data collection (developmental testing, buccal swabs, play-based assessment, questionnaires) will proceed as planned. COSP groups will be conducted remotely via Zoom.
  Interventions: Behavioral: Circle of Security Parenting program
- Waitlist Control Group (No Intervention): This group of mothers will be assigned to a waitlist control group and will be scheduled to begin the parenting skills group at a later time. In order to serve as a no-intervention control, they will be administered assessments while on the waiting list. These assessments will be given concurrently with mid-point assessment of the intervention group.

INTERVENTIONS:
Behavioral: Circle of Security Parenting program — The Circle of Security Parenting (COSP) program is an 8- week group parenting course that was designed using decades of attachment research to foster a secure attachment by teaching parents to read and respond to infant cues, and to recognize the interplay between their own psychological and emotional experiences and the emotional regulation of their infants. The COSP program provides parents with relationship tools and techniques for understanding their children's needs in new ways that provide lasting security for the child and more satisfaction for the parent. There are two major themes in the program: 1) teaching parents how to read their children's behavior and use it as a guide for meeting their needs and 2) helping parents to understand how their own early attachment relationships have influenced them as a person, and how those influences show up in their parenting and impact their ability to help regulate their child and respond to their needs.
  Other Names: COSP
  Arms: Circle of Security Parenting (COSP) group

SUMMARY:
The goal of this longitudinal study is to study the effects of a parenting skills group (Circle of Security Parenting, aka COSP) in mothers with postpartum depression. The main questions it aims to answer are:

* Will changes in methylation of the OXTR rs53576 be apparent in mother and/or infant after having gone through the 8-week COSP program?
* Will COSP participation be associated with improved symptoms of postpartum depression (over and above standard care), attachment style, and relational characteristics of the mother-infant dyad?
* Will COSP participation be associated with changes in social behavior in the infant, and if so, do they persist throughout childhood?

Participants will

* Participate in an 8-week COSP program delivered remotely via Zoom.
* Provide buccal swabs (mother and infant) to assess changes in methylation of OXTR rs53576 pre- versus post-intervention.
* Complete a series of assessment questionnaires delivered remotely.
* Videotape a play-based assessment in their home.
* Receive infant developmental testing

Researchers will compare characteristics of waitlist controls to those participating in the COSP program at the mid-way point of the program to see if the two groups differ.

DETAILED DESCRIPTION:
The primary aims of this study are to 1) better understand the biological/genetic mechanisms and processes of behavior change in mothers and babies relating to oxytocin receptor gene methylation; 2) complete an outcome assessment of the efficacy of the COSP intervention using a tele-health format, specifically in relation to treating maternal depression; 3) to better understand the mechanisms and processes of change in relation to maternal and infant co-regulation achieved through the promotion of a secure attachment between mothers and their at-risk infants, and to understand how these processes form a trajectory of behavioral outcomes in kindergarten.

The COSP program lasts for 8 weeks and will be delivered via Zoom. Researchers will collect a variety of data including biological samples, self-report questionnaires, developmental assessment, and direct observation to assess predictors and outcomes relating to participation in the COSP program. Data will be collected prior to starting COSP, half-way through participation, after having completed the program, and at several timepoints following completion.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged 18-50 years old with infants aged 3-14 months old
* Mothers who are experiencing symptoms of depression and mothers who are not experiencing symptoms of depression (non-depressed controls) are encouraged to participate.

(please note that mothers who are experiencing active depression and who are not already being treated under the care of a qualified healthcare provider (i.e. through therapy or psychopharmacological intervention) will be referred for such treatment prior to being enrolled in the study. This study is not a replacement for professional management of depression or other mental health symptoms.

Exclusion Criteria:

* Mothers with severe psychopathology (such as bipolar disorder, schizophrenia, personality disorders, among others)
* Infants with major medical problems that may interfere with a mother's ability to participate in and benefit from the intervention

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2035-04-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in methylation of OXTR receptor gene rs53576 | Time1 (baseline), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention) Time7 (average 4.5 years post-intervention)
  Buccal swabs from mother and infant
Changes in Beck Depression Inventory, Second Edition (BDI-II) Score | Time1 (baseline), Time2 (1 week pre-intervention), Time3 (week 5 of intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention), Time7 (average 4.5 years post-intervention)
  The BDI-II is a brief, self-report inventory designed to measure the severity of depression symptomatology for ages 13-80 years old and takes approximately 5 minutes to complete. The BDI-II is comprised of 21 items. Each item is scored on a scale of 0 to 3, with a total score range of 0-63. Total score of <14 indicates minimal range, 14-19 indicates mild severity, 20-28 indicates moderate severity, and 29-63 indicates a score in the severe range. Higher scores indicate greater levels of depression.
Changes Postpartum Depression Screening Scale (PDSS) Score | Time1 (baseline), Time2 (1 week pre-intervention), Time3 (week 5 of intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention)
  The PDSS is a 35-item self-report measure helps clinicians identify mothers suffering from postpartum depression. It takes about 5-10 minutes to complete and is written at a third-grade reading level. Mothers respond using a 5-point scale ranging from "strongly disagree" to "strongly agree" and yields an overall severity score. A higher score indicates more severe depression.
Changes in Dyadic Adjustment Scale (DAS) Score | Time1 (baseline), Time2 (1 week pre-intervention), Time3 (week 5 of intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention), Time7 (average 4.5 years post-intervention)
  A 32-item measure of relationship quality. The scale is divided into 4 subscales: (1) Dyadic Consensus - degree to which respondent agrees with partner (2) Dyadic Satisfaction -- degree to which respondent feels satisfied with partner (3) Dyadic Cohesion -degree to which respondent and partner participate in activities together (4) Affectional Expression -degree to which respondent agrees with partner regarding emotional affection. Scores range from 0-151, with higher scores being indicative of more positive dyadic adjustment and lower distress level.

SECONDARY OUTCOMES:
Changes in Denver Maternal Stress Assessment Score | Time1 (baseline), Time2 (1 week pre-intervention), Time3 (week 5 of intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention), Time7 (average 4.5 years post-intervention)
  The Denver Maternal Stress Assessment consists of 13 questions regarding a mothers stress, social support, and health behaviors, along with an inventory of different types of stress encountered in the past year. Results provide qualitative data relating to these categories.
Changes in MacArthur Short Form Vocabulary Checklist Score (child) | Time1 (baseline), Time5 (6 months post-intervention), Time6 (12 months post-intervention)
  The infant short form (Level I, for 8- to 18-month-olds) contains an 89-word checklist for vocabulary comprehension and production.
Changes in Maternal Postnatal Attachment Scale (MPAS) Score | Time1 (baseline), Time2 (1 week pre-intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention)
  The Maternal Postnatal Attachment Scale (MPAS) is a 19 item self-report questionnaire that is used to assess mother-to-infant attachment. According to the authors, parent-to-infant attachment refers to "the emotional bond or tie of affection experienced by the parent towards the infant" (Condon & Corkingdale, 1998). Items are scored on a scale of 1-5, with item totals summed to obtain a scaled score. Lower scores indicate lower attachment and higher scores higher attachment.
Changes in The Multidimensional Scale of Perceived Social Support (MSPSS) Score | Time1 (baseline), Time2 (1 week pre-intervention), Time3 (week 5 of intervention), Time4 (1 week post-intervention), Time5 (6 months post-intervention), Time6 (12 months post-intervention), Time7 (average 4.5 years post-intervention)
  The Multidimensional Scale of Perceived Social Support (Zimet et al., 1988) is a 12-item measure of perceived adequacy of social support from three sources: family, friends, & significant other; using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Changes in Carey Infant Temperament Questionnaire (ITQ) Score | Time1 (baseline), Time5 (6 months post-intervention), Time6 (12 months post-intervention), Time7 (average 4.5 years post-intervention)
  The Carey Temperament Scales are parent report questionnaires that determine behavioral style in each of nine categories of temperament in infants, toddlers, and children up to age 13 years old. Temperament is divided into categories of "easy," "intermediate low" "intermediate high," and "difficult," with lower scores indicating easy temperament and higher indicating more difficult temperament.
Empathy & Theory of Mind Scale (EToMS) Score | Time7 (average 4.5 years post-intervention)
  The Empathy and Theory of Mind Scale (EToMS) is a 17-item measure that was created to assess three specific facets of children's social functioning (empathy, prosocial behaviors that employ theory of mind ability ("Nice" TOM), and antisocial behaviors that employ theory of mind ability ("Nasty" TOM) (Wang & Wang, 2015). This measure was developed to provide an evaluation of children's empathic ability and understanding of epistemic mental states, as well as their prosocial or antisocial behaviors.
Inventory of Callous-Unemotional Traits (ICU) Score | Time7 (average 4.5 years post-intervention)
  The ICU is a 24-item measure that was created to assess three specific facets of affective functioning (callousness, level of care for others, and level of emotionality). These three factors have been shown to differentiate a unique subgroup of individuals who are most at risk for severe antisocial behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Stophaeros, MS, Principal Investigator — sunny.stophaeros@ucdenver.edu
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

REFERENCES:
- [Background] Kendler KS, Karkowski LM, Prescott CA. Causal relationship between stressful life events and the onset of major depression. Am J Psychiatry. 1999 Jun;156(6):837-41. doi: 10.1176/ajp.156.6.837. PMID 10360120
- [Background] Taylor, S. E., & Broffman, J. I. (2011). Psychosocial resources: Functions, origins, and links to mental and physical health. In Advances in experimental social psychology (Vol. 44, pp. 1-57). Academic Press.
- [Background] Taylor, S. E. (2010). Health psychology. Oxford University Press.
- [Background] Moses-Kolko EL, Roth EK. Antepartum and postpartum depression: healthy mom, healthy baby. J Am Med Womens Assoc (1972). 2004 Summer;59(3):181-91. PMID 15354371
- [Background] Darcy JM, Grzywacz JG, Stephens RL, Leng I, Clinch CR, Arcury TA. Maternal depressive symptomatology: 16-month follow-up of infant and maternal health-related quality of life. J Am Board Fam Med. 2011 May-Jun;24(3):249-57. doi: 10.3122/jabfm.2011.03.100201. PMID 21551396
- [Background] Josefsson A, Larsson C, Sydsjo G, Nylander PO. Temperament and character in women with postpartum depression. Arch Womens Ment Health. 2007 Feb;10(1):3-7. doi: 10.1007/s00737-006-0159-3. Epub 2006 Dec 4. PMID 17143777
- [Background] Posmontier B. Functional status outcomes in mothers with and without postpartum depression. J Midwifery Womens Health. 2008 Jul-Aug;53(4):310-8. doi: 10.1016/j.jmwh.2008.02.016. PMID 18586183
- [Background] Cicchetti D, Rogosch FA, Toth SL, Spagnola M. Affect, cognition, and the emergence of self-knowledge in the toddler offspring of depressed mothers. J Exp Child Psychol. 1997 Dec;67(3):338-62. doi: 10.1006/jecp.1997.2412. PMID 9440297
- [Background] Milgrom, J., Westley, D. T., & Gemmill, A. W. (2004). The mediating role of maternal responsiveness in some longer term effects of postnatal depression on infant development. Infant Behavior and Development, 27(4), 443-454.
- [Background] Child care and mother-child interaction in the first 3 years of life. NICHD Early Child Care Research Network. Dev Psychol. 1999 Nov;35(6):1399-413. PMID 10563730
- [Background] Stanley C, Murray L, Stein A. The effect of postnatal depression on mother-infant interaction, infant response to the Still-face perturbation, and performance on an Instrumental Learning task. Dev Psychopathol. 2004 Winter;16(1):1-18. doi: 10.1017/s0954579404044384. PMID 15115062
- [Background] Muzik M, Borovska S. Perinatal depression: implications for child mental health. Ment Health Fam Med. 2010 Dec;7(4):239-47. PMID 22477948
- [Background] Slomian J, Honvo G, Emonts P, Reginster JY, Bruyere O. Consequences of maternal postpartum depression: A systematic review of maternal and infant outcomes. Womens Health (Lond). 2019 Jan-Dec;15:1745506519844044. doi: 10.1177/1745506519844044. PMID 31035856
- [Background] Gentile S. Untreated depression during pregnancy: Short- and long-term effects in offspring. A systematic review. Neuroscience. 2017 Feb 7;342:154-166. doi: 10.1016/j.neuroscience.2015.09.001. Epub 2015 Sep 4. PMID 26343292
- [Background] Garner AS, Shonkoff JP; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. Early childhood adversity, toxic stress, and the role of the pediatrician: translating developmental science into lifelong health. Pediatrics. 2012 Jan;129(1):e224-31. doi: 10.1542/peds.2011-2662. Epub 2011 Dec 26. PMID 22201148
- [Background] Shonkoff JP, Boyce WT, McEwen BS. Neuroscience, molecular biology, and the childhood roots of health disparities: building a new framework for health promotion and disease prevention. JAMA. 2009 Jun 3;301(21):2252-9. doi: 10.1001/jama.2009.754. PMID 19491187
- [Background] Chaudron LH, Szilagyi PG, Campbell AT, Mounts KO, McInerny TK. Legal and ethical considerations: risks and benefits of postpartum depression screening at well-child visits. Pediatrics. 2007 Jan;119(1):123-8. doi: 10.1542/peds.2006-2122. PMID 17200279
- [Background] Kim S, Fonagy P, Koos O, Dorsett K, Strathearn L. Maternal oxytocin response predicts mother-to-infant gaze. Brain Res. 2014 Sep 11;1580:133-42. doi: 10.1016/j.brainres.2013.10.050. Epub 2013 Nov 1. PMID 24184574
- [Background] Breton C, Zingg HH. Expression and region-specific regulation of the oxytocin receptor gene in rat brain. Endocrinology. 1997 May;138(5):1857-62. doi: 10.1210/endo.138.5.5127. PMID 9112379
- [Background] Kimura T, Tanizawa O, Mori K, Brownstein MJ, Okayama H. Structure and expression of a human oxytocin receptor. Nature. 1992 Apr 9;356(6369):526-9. doi: 10.1038/356526a0. PMID 1313946
- [Background] Inoue H, Yamasue H, Tochigi M, Abe O, Liu X, Kawamura Y, Takei K, Suga M, Yamada H, Rogers MA, Aoki S, Sasaki T, Kasai K. Association between the oxytocin receptor gene and amygdalar volume in healthy adults. Biol Psychiatry. 2010 Dec 1;68(11):1066-72. doi: 10.1016/j.biopsych.2010.07.019. Epub 2010 Sep 15. PMID 20832055
- [Background] Tost H, Kolachana B, Hakimi S, Lemaitre H, Verchinski BA, Mattay VS, Weinberger DR, Meyer-Lindenberg A. A common allele in the oxytocin receptor gene (OXTR) impacts prosocial temperament and human hypothalamic-limbic structure and function. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13936-41. doi: 10.1073/pnas.1003296107. Epub 2010 Jul 20. PMID 20647384
- [Background] Furman DJ, Chen MC, Gotlib IH. Variant in oxytocin receptor gene is associated with amygdala volume. Psychoneuroendocrinology. 2011 Jul;36(6):891-7. doi: 10.1016/j.psyneuen.2010.12.004. Epub 2011 Jan 3. PMID 21208749
- [Background] Loth E, Poline JB, Thyreau B, Jia T, Tao C, Lourdusamy A, Stacey D, Cattrell A, Desrivieres S, Ruggeri B, Fritsch V, Banaschewski T, Barker GJ, Bokde AL, Buchel C, Carvalho FM, Conrod PJ, Fauth-Buehler M, Flor H, Gallinat J, Garavan H, Heinz A, Bruehl R, Lawrence C, Mann K, Martinot JL, Nees F, Paus T, Pausova Z, Poustka L, Rietschel M, Smolka M, Struve M, Feng J, Schumann G; IMAGEN Consortium. Oxytocin receptor genotype modulates ventral striatal activity to social cues and response to stressful life events. Biol Psychiatry. 2014 Sep 1;76(5):367-76. doi: 10.1016/j.biopsych.2013.07.043. Epub 2013 Oct 8. PMID 24120094
- [Background] Asherin RM, Everhart KD, Stophaeros SL, Vogeli JM, Fowler J, Phiel CJ, Kaplan PS. Associations between maternal depression and mother and infant oxytocin receptor gene (OXTR_rs53576) polymorphisms. Dev Psychobiol. 2020 May;62(4):496-504. doi: 10.1002/dev.21938. Epub 2019 Nov 21. PMID 31755553
- [Background] Ludmer JA, Gonzalez A, Kennedy J, Masellis M, Meinz P, Atkinson L. Association between maternal childhood maltreatment and mother-infant attachment disorganization: Moderation by maternal oxytocin receptor gene and cortisol secretion. Horm Behav. 2018 Jun;102:23-33. doi: 10.1016/j.yhbeh.2018.04.006. Epub 2018 Apr 24. PMID 29673618
- [Background] Harlow, H. F., & Zimmermann, R. R. (1958). The development of affectional responses in infant monkeys. Proceedings of the American Philosophical Society, 102(5), 501-509.
- [Background] Bell AF, Carter CS, Steer CD, Golding J, Davis JM, Steffen AD, Rubin LH, Lillard TS, Gregory SP, Harris JC, Connelly JJ. Interaction between oxytocin receptor DNA methylation and genotype is associated with risk of postpartum depression in women without depression in pregnancy. Front Genet. 2015 Jul 21;6:243. doi: 10.3389/fgene.2015.00243. eCollection 2015. PMID 26257770
- [Background] Reiner I, Van IJzendoorn MH, Bakermans-Kranenburg MJ, Bleich S, Beutel M, Frieling H. Methylation of the oxytocin receptor gene in clinically depressed patients compared to controls: The role of OXTR rs53576 genotype. J Psychiatr Res. 2015 Jun;65:9-15. doi: 10.1016/j.jpsychires.2015.03.012. Epub 2015 Mar 24. PMID 25890851
- [Background] Unternaehrer E, Luers P, Mill J, Dempster E, Meyer AH, Staehli S, Lieb R, Hellhammer DH, Meinlschmidt G. Dynamic changes in DNA methylation of stress-associated genes (OXTR, BDNF ) after acute psychosocial stress. Transl Psychiatry. 2012 Aug 14;2(8):e150. doi: 10.1038/tp.2012.77. PMID 22892716
- [Background] Bergman Y, Cedar H. DNA methylation dynamics in health and disease. Nat Struct Mol Biol. 2013 Mar;20(3):274-81. doi: 10.1038/nsmb.2518. PMID 23463312
- [Background] Aronica L, Levine AJ, Brennan K, Mi J, Gardner C, Haile RW, Hitchins MP. A systematic review of studies of DNA methylation in the context of a weight loss intervention. Epigenomics. 2017 May;9(5):769-787. doi: 10.2217/epi-2016-0182. PMID 28517981
- [Background] Yaholkoski, A., Hurl, K., & Theule, J. (2016). Efficacy of the circle of security intervention: a meta-analysis. Journal of Infant, Child, and Adolescent Psychotherapy, 15(2), 95-103.
- [Background] Vaever MS, Smith-Nielsen J, Lange T. Copenhagen infant mental health project: study protocol for a randomized controlled trial comparing circle of security -parenting and care as usual as interventions targeting infant mental health risks. BMC Psychol. 2016 Nov 22;4(1):57. doi: 10.1186/s40359-016-0166-8. PMID 27876079
- [Background] Huber A, McMahon CA, Sweller N. EFFICACY OF THE 20-WEEK CIRCLE OF SECURITY INTERVENTION: CHANGES IN CAREGIVER REFLECTIVE FUNCTIONING, REPRESENTATIONS, AND CHILD ATTACHMENT IN AN AUSTRALIAN CLINICAL SAMPLE. Infant Ment Health J. 2015 Nov-Dec;36(6):556-74. doi: 10.1002/imhj.21540. Epub 2015 Nov 9. PMID 26551929